CLINICAL TRIAL: NCT04986579
Title: Assessing the Impact of Scalp Cooling in With Metastatic Breast Cancer
Brief Title: Scalp Cooling in MBC
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Paxman Coolers Limited (Unknown); AstraZeneca (Industry); Eisai Inc. (Industry); Daiichi Sankyo (Industry); Gilead Sciences (Industry)
Responsible Party: Principal Investigator, Elahe Salehi, NP, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 21-169
Record Dates: First submitted 2021-07-20; First posted 2021-08-03 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Metastatic Breast Cancer; Chemotherapy-induced Alopecia
Keywords: Metastatic Breast Cancer; Chemotherapy-induced Alopecia
MeSH Terms: conditions — Breast Neoplasms | interventions — eribulin; sacituzumab govitecan; trastuzumab deruxtecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (6):
- ERIBULIN WITH PAXMAN SCALP COOLING SYSTEM (PSCS) (Experimental): Participants will use Paxman Scalp Cooling System (PSCS) on days 1, 8 and 21 of each of their standard of care (SOC) treatment cycles with Eribulin.
  Study cyle is 21 days with total number of cycles based on discretion of treating provider up to 2 years.
  Interventions: Device: Paxman Scalp Cooling System; Drug: Eribulin
- ERIBULIN WITHOUT PAXMAN SCALP COOLING SYSTEM (PSCS) (Active Comparator): Participants will not use Paxman Scalp Cooling System (PSCS) during their standard of care (SOC) treatment with Eribulin.
  Study cyle is 21 days with total number of cycles based on discretion of treating provider up to 2 years.
  Interventions: Drug: Eribulin
- SACITUZUMAB GOVITECAN WITH PAXMAN SCALP COOLING SYSTEM (PSCS) (Experimental): Participants will use Paxman Scalp Cooling System (PSCS) on days 1 and 21 of each of their standard of care (SOC) treatment cycles with SACITUZUMAB GOVITECAN.
  Study cyle is 21 days with total number of cycles based on discretion of treating provider up to 2 years.
  Interventions: Device: Paxman Scalp Cooling System; Drug: Sacituzumab govitecan
- SACITUZUMAB GOVITECAN WITHOUT PAXMAN SCALP COOLING SYSTEM (PSCS) (Active Comparator): Participants will not use Paxman Scalp Cooling System (PSCS) during their standard of care (SOC) treatment with SACITUZUMAB GOVITECAN.
  Study cyle is 21 days with total number of cycles based on discretion of treating provider up to 2 years.
  Interventions: Drug: Sacituzumab govitecan
- TRASTUZUMAB DERUXTECAN WITH PAXMAN SCALP COOLING SYSTEM (PSCS) (Experimental): Participants will use Paxman Scalp Cooling System (PSCS) on days 1, 8 and 21 of each of their standard of care (SOC) treatment cycles with TRASTUZUMAB DERUXTECAN.
  Study cyle is 21 days with total number of cycles based on discretion of treating provider up to 2 years.
  Interventions: Device: Paxman Scalp Cooling System; Drug: Trastuzumab deruxtecan
- TRASTUZUMAB DERUXTECAN WITHOUT PAXMAN SCALP COOLING SYSTEM (Active Comparator): Participants will not use Paxman Scalp Cooling System (PSCS) during their standard of care (SOC) treatment with TRASTUZUMAB DERUXTECAN.
  Study cyle is 21 days with total number of cycles based on discretion of treating provider up to 2 years.
  Interventions: Drug: Trastuzumab deruxtecan

INTERVENTIONS:
Device: Paxman Scalp Cooling System — Cap attached to coolant lines connected to a refrigeration unit placed on scalp
  Other Names: Scalp Cooling Cap
  Arms: ERIBULIN WITH PAXMAN SCALP COOLING SYSTEM (PSCS); SACITUZUMAB GOVITECAN WITH PAXMAN SCALP COOLING SYSTEM (PSCS); TRASTUZUMAB DERUXTECAN WITH PAXMAN SCALP COOLING SYSTEM (PSCS)
Drug: Eribulin — Intravenous Infusion
  Other Names: Halaven
  Arms: ERIBULIN WITH PAXMAN SCALP COOLING SYSTEM (PSCS); ERIBULIN WITHOUT PAXMAN SCALP COOLING SYSTEM (PSCS)
Drug: Sacituzumab govitecan — Intravenous Infusion
  Other Names: Trodelvy; IMMU-132
  Arms: SACITUZUMAB GOVITECAN WITH PAXMAN SCALP COOLING SYSTEM (PSCS); SACITUZUMAB GOVITECAN WITHOUT PAXMAN SCALP COOLING SYSTEM (PSCS)
Drug: Trastuzumab deruxtecan — Intravenous Infusion
  Other Names: Enhertu; DS-8201a
  Arms: TRASTUZUMAB DERUXTECAN WITH PAXMAN SCALP COOLING SYSTEM (PSCS); TRASTUZUMAB DERUXTECAN WITHOUT PAXMAN SCALP COOLING SYSTEM

SUMMARY:
This research is being done to compare rates of hair loss of people with metastatic breast who use scalp cooling versus those who do not use scalp cooling after receiving standard of care treatment with either sacituzumab govitecan, trastuzumab deruxtecan, or eribulin.

The name of the study intervention involved in this study is:

* Paxman Scalp Cooling System

DETAILED DESCRIPTION:
This study is a prospective, controlled, pivotal clinical investigation to assess the efficacy of the Paxman Scalp Cooling System (PSCS) at preventing hair loss in people undergoing treatment for metastatic breast cancer with either Sacituzumab govitecan (IMMU-132 or Trodelvy™), trastuzumab deruxtecan (DS-8201a or Enhertu®), or Eribulin (Halaven®).

The U.S. Food and Drug Administration (FDA) has approved the Paxman Scalp Cooling System as a treatment option for preventing hair loss while patients are undergoing chemotherapy. This system has however not been specifically studied to look at its ability to prevent hair loss in patients specifically receiving sacituzumab govitecan, trastuzumab deruxtecan, or eribulin.

The research study procedures include: screening for eligibility, photographs, hair loss assessments, questionnaires and study treatment including evaluations and follow up visits.

Participants will receive study treatment with scalp cooling with standard of care chemotherapy treatment and will be followed for 2-4 weeks after completion of treatment with chemotherapy.

It is expected that about 120 people will take part in this research study.

Paxman Coolers Limited is a medical device company and is supporting this research study by providing access to the investigational device, Paxman Scalp Cooling System.

ELIGIBILITY:
Inclusion Criteria:

* Men and women with a diagnosis of metastatic invasive breast cancer with a ECOG PS≤2
* Participant is ≥ 18 years old.
* Hair present at baseline.
* One of the following full dose chemotherapy regimens must be planned for at least 4 cycles:

  * Sacituzumab govitecan (IMMU-132) 10 mg/kg administered intravenously on days 1 and 8 of each 21-day cycle
  * Trastuzumab deruxtecan 5.4 mg/kg administered intravenously once every 3 weeks
  * Eribulin 1.4 mg/m2 administered intravenously on days 1 and 8 of each 21-day cycle
* The Paxman Scalp Cooling System must be initiated with the first dose of therapy in participants that elect to participate in the scalp cooling group.

Exclusion Criteria:

* Known hematological malignancies (i.e. leukemia or lymphoma)
* Known scalp metastases.
* Baseline alopecia (defined CTCAE 5.0 grade > 0, see Appendix B)
* Subjects with cold agglutinin disease or cold urticaria.
* Subjects who are scheduled for bone marrow ablation chemotherapy.
* Personal history of migraines, cluster or tension headaches as defined as actual medical diagnosis by a physician and/ or prescribed medications. If personal history of migraines was related to a past medical problem that is now resolved, the subject may go on study at the discretion of the Principal Investigator.
* Subjects who have lichen planus or lupus.
* Participants who are receiving any additional anti-cancer agents

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2021-10-07 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2028-06-01 (Estimated)

PRIMARY OUTCOMES:
Hair Loss Rate | Up to 2 years
  Hair loss rate defined as CTCAE v5.0 alopecia grade 1 or higher compared in the scalp cooling group using the Paxman Hair Loss Prevention System (PSCS) and group not using scalp cooling.

SECONDARY OUTCOMES:
Change in Patient Reported Quality of Life | Baseline, Day 1 of cycle 3, day 1 of cycle 5, and after completing therapy or at the time of disease progression whichever occurs first up to 2 years. Cycle is 21 days
  The Chemotherapy-Induced Alopecia Distress Scale (CADS) [25] will be used to assess patient reported positive quality of life changes using Paxman Hair Loss Prevention System (PSCS).
Change in Patient Reported Quality of Life | Baseline, Day 1 of cycle 3, day 1 of cycle 5, and after completing therapy or at the time of disease progression whichever occurs first up to 2 years. Cycle is 21 days.
  Body image scale (BIS) will be used to assess patient reported positive quality of life changes using Paxman Hair Loss Prevention System (PSCS).

CONTACTS AND LOCATIONS:
Overall Officials: Elahe Salehi, DNP, ANP-BC, Principal Investigator — Dana-Farber Cancer Institute
Locations (2):
- United States (2):
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to: [contact information for Sponsor Investigator or designee]. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: Contact the Belfer Office for Dana-Farber Innovations (BODFI) at innovation@dfci.harvard.edu